CLINICAL TRIAL: NCT04446117
Title: A Phase 3, Randomized, Open-Label, Controlled Study of Cabozantinib (XL184) in Combination With Atezolizumab vs Second Novel Hormonal Therapy (NHT) in Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of Cabozantinib in Combination With Atezolizumab Versus Second NHT in Subjects With mCRPC
Acronym: CONTACT-02
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Collaborators: Roche-Genentech (Industry); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-315
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Prostate Cancer; Prostate Adenocarcinoma
Keywords: prostate cancer; castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib; atezolizumab; Abiraterone Acetate; abiraterone; enzalutamide; Prednisone

STUDY DESIGN:
Intervention Model Description: Approximately 580 eligible subjects will be randomized in a 1:1 fashion to the experimental arm receiving cabozantinib and atezolizumab in combination (290) or to the control arm receiving a second NHT (290).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Subjects with mCRPC will receive cabozantinib 40mg oral, qd + atezolizumab 1200mg infusion, q3w
  Interventions: Drug: Cabozantinib; Drug: Atezolizumab
- Control Arm (Active Comparator): Subjects with mCRPC will receive active comparator of EITHER abiraterone 1000mg oral, qd + prednisone 5 mg oral, bid; OR enzalutamide 160mg oral, qd as designated by the Investigator prior to randomization
  Interventions: Drug: Abiraterone Acetate; Drug: Enzalutamide; Drug: Prednisone

INTERVENTIONS:
Drug: Cabozantinib — Supplied as 20-mg tablets; administered orally daily at 40mg
  Other Names: XL184; Cabometyx®
  Arms: Experimental Arm
Drug: Atezolizumab — Supplied as 1200 mg/20 mL vials; administered as an IV infusion once every 3 weeks (q3w)
  Other Names: Tecentriq®
  Arms: Experimental Arm
Drug: Abiraterone Acetate — Supplied as 500 mg tablets; administered orally daily at 1000mg with prednisone 5 mg orally bid
  Other Names: Abiraterone; Zytiga
  Arms: Control Arm
Drug: Enzalutamide — Supplied as 40 mg capsules; administered orally daily at 160mg
  Other Names: Xtandi
  Arms: Control Arm
Drug: Prednisone — Supplied as 5 mg tablets; administered orally bid at 5 mg with abiraterone 1000mg orally daily
  Arms: Control Arm

SUMMARY:
This is a Phase 3, multi-center, randomized, open-label, controlled study designed to evaluate the safety and efficacy of cabozantinib given in combination with atezolizumab versus a second novel hormonal therapy (NHT) in men with metastatic castration-resistant prostate cancer (mCRPC) who have previously been treated with one, and only one, NHT for their prostate cancer disease.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of cabozantinib (XL184) in combination with atezolizumab versus a second NHT (abiraterone or enzalutamide) in subjects with mCRPC who have previously been treated with one, and only one, NHT (e.g. abiraterone, apalutamide, darolutamide, or enzalutamide) to treat metastatic castration-sensitive prostate cancer (mCSPC), non-metastatic CRPC (M0 CRPC), or mCRPC, and who have measurable extrapelvic disease. The multiple primary efficacy endpoints comparing the experimental arm and control arm are Duration of Progression Free Survival (PFS) per RECIST 1.1 by Blinded Independent Radiology Committee (BIRC) and Duration of Overall Survival (OS). The secondary efficacy endpoint is Objective Response Rate (ORR) per RECIST 1.1 per BIRC.

ELIGIBILITY:
Inclusion Criteria:

* Men with histologically or cytologically confirmed adenocarcinoma of the prostate
* Prior treatment with one, and only one, NHT (eg, abiraterone, apalutamide, darolutamide, or enzalutamide) for castration-sensitive locally advanced (T3 or T4) or mCSPC, M0 CRPC, or mCRPC
* Surgical or medical castration, with serum testosterone ≤ 50 ng/dL (≤ 1.73 nmol/L) at screening
* Measurable (extrapelvic soft tissue) metastatic disease per Investigator assessment defined by at least one of the following: measurable visceral disease (eg, adrenal, kidney, liver, lung, pancreas, spleen) per RECIST 1.1; OR measurable extrapelvic adenopathy (ie, adenopathy above the aortic bifurcation)
* Progressive disease at study entry as defined by specific criteria for prostate specific antigen (PSA) progression OR soft tissue disease progression in the opinion of the Investigator (Note: subjects with bone disease progression alone are not eligible)
* Age ≥ 18 years old or meeting country definition of adult, whichever is older, on the day of consent
* ECOG performance status of 0 or 1
* Recovery to baseline or ≤ Grade 1 per Common Terminology Criteria for Adverse Events (CTCAE) v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy in the opinion of the Investigator
* Adequate organ and marrow function based upon specific laboratory assessments obtained within 21 days prior to randomization
* Understanding and ability to comply with protocol requirements

Exclusion Criteria:

* Any prior nonhormonal therapy initiated for the treatment of mCRPC
* Receipt of abiraterone within 1 week; cyproterone within 10 days; or flutamide, nilutamide, bicalutamide, enzalutamide, or other androgen-receptor inhibitors within 2 weeks before randomization
* Radiation therapy within 4 weeks (2 weeks for bone metastases) prior to randomization (subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible)
* Known brain metastases or cranial epidural disease unless adequately treated and clinically stable at least 4 weeks prior to randomization
* Symptomatic or impending spinal cord compression or cauda equina syndrome
* Concomitant anticoagulation with oral anticoagulants (some specific exceptions apply)
* Administration of a live, attenuated vaccine within 30 days prior to randomization
* Systematic treatment with, or any condition requiring, either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to randomization
* Uncontrolled, significant intercurrent or recent illness
* Major surgery within 4 weeks prior to randomization
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms per ECG within 21 days before randomization
* Inability or unwillingness to swallow pills or receive IV administration
* Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies
* Any other active malignancy at time of randomization or diagnosis of another malignancy within 2 years prior to randomization that requires active treatment (some exceptions apply such as locally curable cancers that have apparently been cured).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2026-10-16 (Estimated)

CONTACTS AND LOCATIONS:
Locations (280):
- United States (36):
  - Exelixis Clinical Site #4, Tucson, Arizona
  - Exelixis Clinical Site #42, Duarte, California
  - Exelixis Clinical Site #2, Fullerton, California
  - Exelixis Clinical Site #224, La Jolla, California
  - Exelixis Clinical Site #3, Marina del Rey, California
  - Exelixis Clinical Site #114, San Diego, California
  - Exelixis Clinical Site #125, Santa Monica, California
  - Exelixis Clinical Site #245, Stanford, California
  - Exelixis Clinical Site #91, Aurora, Colorado
  - Exelixis Clinical Site #14, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Yale University, School of Medicine, New Haven, Connecticut
  - Exelixis Clinical Site #108, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Exelixis Clinical Site #215, Westwood, Kansas
  - Exelixis Clinical Site #242, Louisville, Kentucky
  - Exelixis Clinical Site #6, Baltimore, Maryland
  - Non-participating Site, Detroit, Michigan
  - Exelixis Clinical Site #203, Rochester, Minnesota
  - Exelixis Clinical Site #19, Omaha, Nebraska
  - Exelixis Clinical Site #144, Las Vegas, Nevada
  - Exelixis Clinical Site #123, East Brunswick, New Jersey
  - Non-participating Site, Lawrenceville, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Exelixis Clinical Site #198, The Bronx, New York
  - Exelixis Site #159, Cleveland, Ohio
  - Exelixis Clinical Site #221, Oklahoma City, Oklahoma
  - Exelixis Clinical Site #18, Philadelphia, Pennsylvania
  - Exelixis Clinical Site #201, Pittsburgh, Pennsylvania
  - Exelixis Clinical Site #1, Nashville, Tennessee
  - Exelixis Clinical Site #5, Houston, Texas
  - Exelixis Clinical Site #177, Houston, Texas
  - Exelixis Clinical Site #259, Houston, Texas
  - Exelixis Clinical Site #41, Temple, Texas
  - Exelixis Clinical Site #67, Salt Lake City, Utah
  - Exelixis Clinical Site #143, Roanoke, Virginia
- Argentina (13):
  - Exelixis Clinical Site #122, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Exelixis Clinical Site #120, Mar del Plata, Buenos Aires
  - Exelixis Site #170, Pergamino, Buenos Aires
  - Exelixis Clinical Site #210, Córdoba, Córdoba Province
  - Exelixis Clinical Site #152, Viedma, Río Negro Province
  - Exelixis Clinical Site #183, Rosario, Santa Fe Province
  - Exelixis Clinical #261, Rosario, Santa Fe Province
  - Exelixis Clinical Site #200, Buenos Aires
  - Exelixis Clinical Site #256, Caba
  - Exelixis Clinical Site #44, Ciudad Autonoma de Buenos Aire
  - Exelixis Clinical Site #105, La Rioja
  - Exelixis Clinical Site #124, San Juan
  - Exelixis Clinical Site #101, San Salvador de Jujuy
- Australia (14):
  - Exelixis Clinical Site #151, Garran, Australian Capital Territory
  - Exelixis Clinical Site #252, Port Macquarie, New South Wales
  - Exelixis Clinical Site #175, Saint Leonards, New South Wales
  - Exelixis Clinical Site # 189, Sydney, New South Wales
  - Exelixis Site #162, Wollongong, New South Wales
  - Exelixis Clinical Site #253, Chermside, Queensland
  - Exelixis Clinical Site #103, Launceston, Tasmania
  - Exelixis Clinical Site #79, Ballarat, Victoria
  - Exelixis Clinical Site #95, Frankston, Victoria
  - Exelixis Clinical #262, Geelong, Victoria
  - Exelixis Clinical Site #53, Melbourne, Victoria
  - Exelixis Clinical Stie #260, Saint Albans, Victoria
  - Exelixis Clinical Site #115, Adelaide
  - Exelixis Clinical Site #149, Box Hill
- Austria (3):
  - Exelixis Clinical Site #156, Linz, Upper Austria
  - Exelixis Site #158, Linz, Upper Austria
  - Exelixis Clinical Site #218, Vienna
- Belgium (4):
  - Exelixis Clinical Site #126, Bonheiden, Antwerpen
  - Exelixis Clinical Site #39, Ghent, Oost-Vlaanderen
  - Exelixis Clinical Site #141, Brussels
  - Exelixis Site #165, Roeselare
- Brazil (14):
  - Exelixis Site #163, Curitiba, Paraná
  - Exelixis Clinical Site #204, Curitiba, Paraná
  - Exelixis Clinical Site #171, Rio de Janeiro, Rio de Janeiro
  - Exelixis Site #157, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #132, Blumenau, Santa Catarina
  - Exelixis Clinical Site #191, Campinas, São Paulo
  - Exelixis Clinical Site #128, Ribeirão Preto, São Paulo
  - Exelixis Clinical Site #106, São José do Rio Preto, São Paulo
  - Exelixis Site #161, São Paulo, São Paulo
  - Exelixis Clinical Site #154, Barretos
  - Exelixis Clinical Site #140, Fortaleza
  - Exelixis Clinical Site #153, Porto Alegre
  - Exelixis Clinical Site #145, Ribeirão Preto
  - Exelixis Clinical Site #116, Santa Cruz do Sul
- Canada (8):
  - Exelixis Clinical Site #69, Edmonton, Alberta
  - Exelixis Clinical Site #112, Kelowna, British Columbia
  - Exelixis Clinical Site #147, Moncton, New Brunswick
  - Exelixis Clinical Site #83, Hamilton, Ontario
  - Exelixis Clinical Site #127, London, Ontario
  - Exelixis Clinical Site #7, Oakville, Ontario
  - Exelixis Clinical Site #178, Granby, Quebec
  - Exelixis Site #160, Montreal, Quebec
- Chile (8):
  - Exelixis Clinical Site #247, Viña del Mar, Región de Valparaíso
  - Exelixis Clinical #263, Santiago, Santiago Metropolitan
  - Exelixis Clinical Site #139, Santiago, Santiago Metropolitan
  - Exelixis Clinical Site #142, Providencia
  - Exelixis Clinical Site #148, Recoleta
  - Exelixis Clinical Site #90, Santiago
  - Exelixis Clinical Site #113, Temuco
  - Exelixis Clinical Site #119, Valparaíso
- Czechia (6):
  - Exelixis Clinical Site #63, Prague, Prague
  - Exelixis Clinical Site #129, Brno
  - Exelixis Clinical Site #130, Olomouc
  - Exelixis Clinical Site #80, Prague
  - Exelixis Clinical Site #31, Prague
  - Exelixis Clinical Site #47, Prague
- France (15):
  - Exelixis Clinical Site #134, Brest
  - Exelixis Clinical Site #77, Clermont-Ferrand
  - Exelixis Clinical Site #155, Dijon
  - Exelixis Clinical Site #74, Hyères
  - Exelixis Clinical Site #222, La Roche-sur-Yon
  - Exelixis Clinical Site #146, Nîmes
  - Exelixis Clinical Site #38, Paris
  - Exelixis Clinical Site #66, Quimper
  - Exelixis Clinical Site #214, Reims
  - Exelixis Clinical Site #135, Saint-Grégoire
  - Exelixis Clinical Site #213, Strasbourg
  - Exelixis Clinical Site #36, Strasbourg
  - Exelixis Clinical Site #73, Toulouse
  - Exelixis Clinical Site #85, Toulouse
  - Exelixis Clinical Site #230, Vandœuvre-lès-Nancy
- Georgia (6):
  - Exelixis Clinical Site #16, Tbilisi
  - Exelixis Clinical Site #9, Tbilisi
  - Exelixis Clinical Site #10, Tbilisi
  - Exelixis Clinical Site #11, Tbilisi
  - Exelixis Clinical Site #15, Tbilisi
  - Exelixis Clinical Site #8, Tbilisi
- Germany (9):
  - Exelixis Clinical Site #176, Nürtingen, Baden-Wurttemberg
  - Exelixis Clinical Site #180, Duisburg, North Rhine-Westphalia
  - Exelixis Clinical Site #98, Gütersloh, North Rhine-Westphalia
  - Exelixis Clinical Site #179, Münster, North Rhine-Westphalia
  - Exelixis Clinical Site #185, Lübeck, Schleswig-Holstein
  - Exelixis Clinical Site #227, Berlin
  - Exelixis Clinical Site #239, Hamburg
  - Exelixis Clinical Site #273, Hanover
  - Exelixis Clinical Site #136, Tübingen
- Greece (9):
  - Exelixis Clinical Site #238, Athens, Attica
  - Exelixis Clinical Site #93, Cholargós, Attica
  - Exelixis Clinical Site #202, Marousi, Attica
  - Exelixis Clinical Site #92, Marousi, Attica
  - Exelixis Clinical Site #244, Nea Kifissia, Attica
  - Exelixis Clinical Site #99, Neo Faliro, Attica
  - Exelixis Clinical Site #45, Heraklion, Crete
  - Exelixis Clinical Site #64, Thessaloniki, Macedonia
  - Exelixis Clinical Site #97, Larissa, Thessaly
- Hungary (6):
  - Exelixis Clinical Site #118, Budapest
  - Exelixis Clinical Site #207, Budapest
  - Exelixis Clinical Site #57, Budapest
  - Exelixis Clinical Site #109, Budapest
  - Exelixis Clinical Site #240, Debrecen
  - Exelixis site #167, Gyula
- Israel (6):
  - Exelixis Clinical Site #55, Haifa
  - Exelixis Clinical Site #27, Jerusalem
  - Exelixis Clinical Site #150, Petah Tikva
  - Exelixis Clinical Site #117, Ramat Gan
  - Exelixis Clinical Site #30, Safed
  - Exelixis Clinical Site #35, Tel Aviv
- Italy (15):
  - Exelixis Site #168, Meldola, FC
  - Exelixis Clinical Site #246, Rozzano, Milano
  - Exelixis Site #156, Sondrio, SO
  - Exelixis Clinical Site #199, Trento, Trentino-Alto Adige
  - Exelixis Clinical Site #217, Ancona
  - Exelixis Clinical Site #121, Florence
  - Exelixis Clinical Site #192, Milan
  - Exelixis Clinical Site #258, Milan
  - Exelixis Clinical #267, Parma
  - Exelixis Clinical Site #237, Pavia
  - Exelixis Clinical Site #107, Perugia
  - Exelixis Clinical #269, Pisa
  - Exelixis Clinical Site #62, Roma
  - Exelixis Clinical Site #234, Roma
  - Exelixis Clinical Site #96, Terni
- Japan (24):
  - Exelixis Clinical Site #232, Toyota-shi, Aichi-ken
  - Exelixis Clinical Site #100, Akita, Akita
  - Exelixis Clinical Site #104, Hirosaki, Aomori
  - Exelixis Clinical Site #43, Kashiwa-shi, Chiba
  - Exelixis Clinical Site #54, Sakura-shi, Chiba
  - Exelixis Clinical Site #72, Sapporo, Hokkaido
  - Exelixis Clinical Site #37, Sapporo, Hokkaido
  - Exelixis Clinical Site #70, Kobe, Hyōgo
  - Exelixis Clinical Site #52, Kobe, Hyōgo
  - Exelixis Clinical Site #84, Kita-gun, Kagawa-ken
  - Exelixis Clinical Site #68, Sagamihara, Kanagawa
  - Exelixis Clinical Site #22, Yokohama, Kanagawa
  - Exelixis Clinical Site #211, Natori-shi, Miyagi
  - Exelixis Clinical Site #88, Chūōku, Osaka-shi
  - Exelixis Clinical Site #51, Hidaka, Saitama
  - Exelixis Clinical Site #216, Shizuoka, Shizuoka
  - Exelixis Clinical Site #65, Shinjuku-Ku, Tokyo
  - Exelixis Clinical Site #61, Ube, Yamaguchi
  - Exelixis Clinical Site #78, Chiba
  - Exelixis Clinical Site #209, Fukuoka
  - Exelixis Clinical Site #26, Nagano
  - Exelixis Clinical Site #81, Ōsaka-sayama
  - Exelixis Clinical Site #75, Tokyo
  - Exelixis Clinical Site #32, Wakayama
- Mexico (14):
  - Exelixis Clinical Site #206, Tuxtla Gutiérrez, Chiapas
  - Exelixis Clinical Site #254, León, Guanajuato
  - Exelixis Clinical Site #212, Guadalajara, Jalisco
  - Exelixis Clinical Site #173, Guadalajara, Jalisco
  - Exelixis Clinical Site #219, Zapopan, Jalisco
  - Exelixis Clinical Site #187, Mexico City, Mexico City
  - Exelixis Clinical Site #257, Monterrey, Nuevo León
  - Exelixis Clinical Site #172, Querétaro City, Querétaro
  - Exelixis Clinical Site #182, Querétaro City, Querétaro
  - Exelixis Clinical Site #250, San Luis Potosí City, San Luis Potosí
  - Exelixis Clinical Site #184, San Luis Potosí City, San Luis Potosí
  - Exelixis Clinical Site #208, Culiacán, Sinaloa
  - Exelixis Clinical Site #174, Mexico City
  - Exelixis Clinical Site #272, Puebla City
- Poland (4):
  - Exelixis Clinical Site #243, Otwock, Masovian Voivodeship
  - Exelixis Clinical Site #82, Bydgoszcz
  - Exelixis Clinical #268, Lodz
  - Exelixis Clinical Site #89, Poznan
- Portugal (8):
  - Exelixis Clinical Site #110, Braga
  - Exelixis Clinical Site #188, Guimarães
  - Exelixis Site #164, Lisbon
  - Exelixis Clinical Site #197, Lisbon
  - Exelixis Clinical Site #196, Loures
  - Exelixis Clinical Site #56, Porto
  - Exelixis Clinical Site #223, Porto
  - Exelixis Clinical Site #193, Vila Real
- Russia (3):
  - Exelixis Site #166, Moscow
  - Exelixis Clinical Site #137, Saint Petersburg
  - Exelixis Clinical Site #195, Saint Petersburg
- Singapore (3):
  - Exelixis Clinical Site #50, Singapore
  - Exelixis Clinical Site #87, Singapore
  - Exelixis Clinical Site #181, Singapore
- South Korea (13):
  - Exelixis Clinical Site #20, Junggu, Daejeon
  - Exelixis Clinical Site #49, Goyang-si, Gyeonggi-do
  - Exelixis Clinical Site #60, Seongnam-si, Gyeonggi-do
  - Exelixis Clinical Site #34, Hwasun, Jeollanam-do
  - Exelixis Clinical Site #58, Busan
  - Exelixis Clinical Site #24, Busan
  - Exelixis Clinical Site #94, Daegu
  - Exelixis Clinical Site #21, Daegu
  - Exelixis Clinical Site #40, Gwangju
  - Exelixis Clinical Site #59, Seoul
  - Exelixis Clinical Site #46, Seoul
  - Exelixis Clinical Site #25, Seoul
  - Exelixis Clinical Site #48, Seoul
- Spain (21):
  - Exelixis Clinical Site #229, Elche, Alicante
  - Exelixis Clinical Site #220, Palma de Mallorca, Balearic Islands
  - Exelixis Clinical Site #12, Manresa, Barcelona
  - Exelixis Clinical Site #233, Santiago de Compostela, La Coruna
  - Exelixis Clinical Site #17, Alcorcón, Madrid
  - Exelixis Clinical Site #225, Oviedo, Principality of Asturias
  - Exelixis Clinical Site #274, Badalona
  - Exelixis Clinical Site #228, Barcelona
  - Exelixis Clinical Site #23, Barcelona
  - Exelixis Clinical Site #255, Barcelona
  - Exelixis Clinical Site #190, Barcelona
  - Exelixis Clinical Site #226, Cadiz
  - Exelixis Clinical Site #33, Córdoba
  - Exelixis Clinical Site #28, Lugo
  - Exelixis Clinical Site #131, Madrid
  - Exelixis Clinical Site #248, Madrid
  - Exelixis Clinical Site #236, Madrid
  - Exelixis Clinical Site #251, Madrid
  - Exelixis Clinical Site #13, Madrid
  - Exelixis Clinical #270, Málaga
  - Exelixis Clinical Site #29, Seville
- Taiwan (8):
  - Exelixis Clinical #266, Kaohsiung City
  - Exelixis Clinical Site #138, Kaohsiung City
  - Exelixis Clinical Site #86, Taichung
  - Exelixis Clinical Site #133, Taichung
  - Exelixis Clinical Site #111, Tainan
  - Exelixis Clinical Site #271, Tainan
  - Exelixis Clinical #264, Taipei
  - Exelixis Clinical #265, Taoyuan District
- Ukraine (4):
  - Exelixis Clinical Site #102, Dnipro
  - Exelixis Clinical Site #186, Dnipro
  - Exelixis Clinical Site #76, Kyiv
  - Exelixis Clinical Site #71, Lutsk
- United Kingdom (6):
  - Exelixis Clinical Site #205, London, England
  - Exelixis Clinical Site #235, Surrey Quays, England
  - Exelixis Clinical Site #241, Taunton, England
  - Exelixis Clinical Site #249, Blackburn, Lancashire
  - Exelixis Clinical Site #231, Northwood, Middlesex
  - Exelixis Clinical Site #194, Swansea, Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal N, Azad AA, Carles J, Matsubara N, Oudard S, Saad F, Merseburger AS, Soares A, McGregor BA, Zurawski B, Tsiatas M, North S, Bondarenko I, Alfie M, Bournakis E, Antonuzzo L, Evilevitch L, Simmons A, Wang F, Ferraldeschi R, Nandoskar P, Pal SK. Cabozantinib plus atezolizumab in metastatic prostate cancer (CONTACT-02): final analyses from a phase 3, open-label, randomised trial. Lancet Oncol. 2025 Jul;26(7):860-876. doi: 10.1016/S1470-2045(25)00209-8. Epub 2025 Jun 13. PMID 40523369
- [Derived] Agarwal N, Azad A, Carles J, Chowdhury S, McGregor B, Merseburger AS, Oudard S, Saad F, Soares A, Benzaghou F, Kerloeguen Y, Kimura A, Mohamed N, Panneerselvam A, Wang F, Pal S. A phase III, randomized, open-label study (CONTACT-02) of cabozantinib plus atezolizumab versus second novel hormone therapy in patients with metastatic castration-resistant prostate cancer. Future Oncol. 2022 Mar;18(10):1185-1198. doi: 10.2217/fon-2021-1096. Epub 2022 Jan 17. PMID 35034502

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study is ongoing, so the results reported are based on a data cutoff date of 19 April 2024.
Groups:
- Experimental Arm: Cabozantinib and Atezolizumab: Participants with metastatic castration-resistant prostate cancer (mCRPC) received cabozantinib 40 milligrams (mg) as oral tablets once daily (QD) throughout the treatment period. Participants also received atezolizumab 1200 mg as an intravenous (IV) infusion once every 3 weeks, administered on Day 1 of each 21-day cycle throughout the treatment period.
  Participants received study treatment as long as they continued to experience clinical benefit in the opinion of the Investigator or until there was unacceptable toxicity, the need for subsequent systemic anticancer treatment, or any other reasons for the treatment discontinuation.
- Control Arm: Second Novel Hormonal Therapy (NHT): Participants with mCRPC received either abiraterone 1000 mg as oral tablets QD and prednisone 5 mg as oral tablets twice daily (BID) or enzalutamide 160 mg as oral tablets QD throughout the treatment period. Participants received study treatment as long as they continued to experience clinical benefit in the opinion of the Investigator or until there was unacceptable toxicity, the need for subsequent systemic anticancer treatment, or any other reasons for the treatment discontinuation.
Period: Overall Study
Arm/Group | Experimental Arm: Cabozantinib and Atezolizumab | Control Arm: Second Novel Hormonal Therapy (NHT)
Started | 289 | 286
Received at Least 1 Dose of Any Study Treatment | 284 | 284
Received Cabozantinib or Atezolizumab | 284 | 0
Received Abiraterone and Prednisone or Enzalutamide (One participant randomized to the experimental arm received a second NHT in error.) | 1 | 283
Discontinued Radiographic Follow-up | 267 | 265
Discontinued Survival Follow-up | 202 | 202
Completed (Participants not completed refers to the number of participants who discontinued from cabozantinib, abiraterone or enzalutamide. 'Completed' refers to the number of participants who were on any study treatment (cabozantinib, atezolizumab, abiraterone or enzalutamide) at the time of data cutoff.) | 22 | 20
Not Completed | 267 | 266
Not completed — No Study Treatment Given | 4 | 3
Not completed — Radiographic Disease Progression | 132 | 158
Not completed — Adverse Event | 79 | 43
Not completed — Lack of Clinical Benefit | 1 | 1
Not completed — Withdrawal by Subject | 24 | 22
Not completed — Lost to Follow-up | 0 | 3
Not completed — Miscellaneous | 26 | 36
Not completed — Missing Data/Data not yet Received | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: Included all participants who were randomized regardless of whether any study treatment or the correct study treatment was received.
Groups:
- Experimental Arm: Cabozantinib and Atezolizumab: Participants with mCRPC received cabozantinib 40 mg as oral tablets QD throughout the treatment period. Participants also received atezolizumab 1200 mg as an IV infusion once every 3 weeks, administered on Day 1 of each 21-day cycle throughout the treatment period.
  Participants received study treatment as long as they continued to experience clinical benefit in the opinion of the Investigator or until there was unacceptable toxicity, the need for subsequent systemic anticancer treatment, or any other reasons for the treatment discontinuation.
- Control Arm: Second NHT: Participants with mCRPC received either abiraterone 1000 mg as oral tablets QD and prednisone 5 mg as oral tablets BID or enzalutamide 160 mg as oral tablets QD throughout the treatment period. Participants received study treatment as long as they continued to experience clinical benefit in the opinion of the Investigator or until there was unacceptable toxicity, the need for subsequent systemic anticancer treatment, or any other reasons for the treatment discontinuation.
- Total: Total of all reporting groups
Arm/Group | Experimental Arm: Cabozantinib and Atezolizumab | Control Arm: Second NHT | Total
Number analyzed (Participants) | 289 | 286 | 575
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 67 | 121
  >=65 years | 235 | 219 | 454
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 289 | 286 | 575
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 72 | 149
  Not Hispanic or Latino | 196 | 196 | 392
  Unknown or Not Reported | 16 | 18 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 3 | 9 | 12
  Asian | 39 | 39 | 78
  Black/African American | 0 | 9 | 9
  Native Hawaiian/Pacific Islander | 1 | 0 | 1
  White | 227 | 213 | 440
  Multiple | 1 | 0 | 1
  Other | 2 | 3 | 5
  Not Reported | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Duration of Progression Free Survival (PFS) Per Response Evaluable Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Radiology Committee (BIRC)
Description: Duration of PFS was defined as the time from randomization to the earlier of either the date of radiographic progression (defined as progressive disease [PD] per RECIST 1.1) per BIRC or the date of death due to any cause. PD was defined as at least a 20% increase in the sum of diameters of target lesions, with an absolute increase of ≥ 5 mm, unequivocal progression of non-target lesions and/or the appearance of new lesions.
Time Frame: Up to a maximum of approximately 30 months (Median duration of follow-up was 14.31 months)
Population: PFS ITT (PITT) analysis population: Included the first 400 participants who were randomized to the Experimental Arm or Control Arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm: Cabozantinib and Atezolizumab | Control Arm: Second NHT
Number analyzed (Participants) | 200 | 200
months | 6.34 [6.18 to 8.80] | 4.17 [3.71 to 5.65]
Statistical Analysis 1: Comparison: Experimental Arm: Cabozantinib and Atezolizumab vs Control Arm: Second NHT; Test type: Superiority; p = 0.0007, Log Rank — Stratification factors used: Liver metastasis, prior docetaxel use for locally advanced or metastatic castration-sensitive prostate cancer (mCSPC) and disease state at first NHT; Cox Proportional Hazard = 0.65, 95% CI 2-sided [0.50 to 0.84] — Stratification factors used: Liver metastasis, prior docetaxel use for locally advanced or mCSPC and disease state at first NHT

2. Primary Outcome: Duration of Overall Survival (OS)
Description: Duration of OS was defined as the time from randomization to death due to any cause. For participants, who were not known to have died at the time of data cutoff and were permanently lost to follow-up, duration of OS was censored at the earlier of the following dates: date the participant was last known to be alive or date of full withdrawal of consent (including survival follow-up), or date of data cutoff.
  OS was calculated as earlier of date of death or censoring - date of randomization + 1)/30.4375
Time Frame: Up to a maximum of approximately 45 months (Median duration of follow-up was 24.05 months)
Population: ITT population: Included all participants who were randomized regardless of whether any study treatment or the correct study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm: Cabozantinib and Atezolizumab | Control Arm: Second NHT
Number analyzed (Participants) | 289 | 286
months | 14.78 [13.37 to 16.66] | 14.98 [13.01 to 18.50]
Statistical Analysis 1: Comparison: Experimental Arm: Cabozantinib and Atezolizumab vs Control Arm: Second NHT; Test type: Superiority; p = 0.2956, Log Rank — Stratification factors used: Liver metastasis, prior docetaxel use for locally advanced or mCSPC and disease state at first NHT; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.72 to 1.10]

ADVERSE EVENTS:
Time Frame: Up to a maximum of approximately 45 months
Description: Safety Population: Consisted of all participants who received any amount of study treatment. Participants were analyzed according to the actual treatment received.
Arm/Group | Experimental Arm: Cabozantinib and Atezolizumab | Control Arm: Second NHT
All-Cause Mortality (participants affected / at risk) | 173/284 | 179/284
Serious Adverse Events (participants affected / at risk) | 135/284 | 89/284
Other Adverse Events (participants affected / at risk) | 281/284 | 254/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm: Cabozantinib and Atezolizumab (N=284) | Control Arm: Second NHT (N=284)
Pneumonia (Infections and infestations) | 8 | 2
Urinary tract infection (Infections and infestations) | 7 | 4
Anal abscess (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 2
Urosepsis (Infections and infestations) | 2 | 1
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Emphysematous cystitis (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 2
Soft tissue infection (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Urinary tract abscess (Infections and infestations) | 1 | 0
Urinary tract candidiasis (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pulmonary sepsis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 20
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour hyperprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 9 | 3
Urinary retention (Renal and urinary disorders) | 8 | 1
Haematuria (Renal and urinary disorders) | 2 | 4
Hydronephrosis (Renal and urinary disorders) | 2 | 2
Urinary tract obstruction (Renal and urinary disorders) | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Bladder perforation (Renal and urinary disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 5 | 3
Pyrexia (General disorders) | 4 | 1
General physical health deterioration (General disorders) | 3 | 6
Oedema peripheral (General disorders) | 3 | 2
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Prosthetic cardiac valve thrombosis (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Pain (General disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Immune-mediated encephalitis (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Anomalous atrioventricular excitation (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0
Arteritis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 2 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Autoimmune thyroid disorder (Endocrine disorders) | 1 | 0
Immune-mediated adrenal insufficiency (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Primary adrenal insufficiency (Endocrine disorders) | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm: Cabozantinib and Atezolizumab (N=284) | Control Arm: Second NHT (N=284)
Diarrhoea (Gastrointestinal disorders) | 133 | 19
Stomatitis (Gastrointestinal disorders) | 56 | 3
Nausea (Gastrointestinal disorders) | 80 | 36
Abdominal pain (Gastrointestinal disorders) | 35 | 10
Constipation (Gastrointestinal disorders) | 48 | 27
Vomiting (Gastrointestinal disorders) | 35 | 17
Dry mouth (Gastrointestinal disorders) | 16 | 0
Dyspepsia (Gastrointestinal disorders) | 16 | 1
Alanine aminotransferase increased (Investigations) | 69 | 9
Aspartate aminotransferase increased (Investigations) | 70 | 15
Weight decreased (Investigations) | 55 | 14
Blood thyroid stimulating hormone increased (Investigations) | 21 | 2
Blood lactate dehydrogenase increased (Investigations) | 21 | 6
Lipase increased (Investigations) | 21 | 7
Gamma-glutamyltransferase increased (Investigations) | 19 | 7
Amylase increased (Investigations) | 16 | 5
Blood alkaline phosphatase increased (Investigations) | 16 | 14
Blood creatinine increased (Investigations) | 15 | 17
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 47 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 5
Rash (Skin and subcutaneous tissue disorders) | 17 | 7
Hypothyroidism (Endocrine disorders) | 65 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 39 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 17
Asthenia (General disorders) | 77 | 37
Fatigue (General disorders) | 85 | 57
Pyrexia (General disorders) | 34 | 9
Oedema peripheral (General disorders) | 23 | 21
Decreased appetite (Metabolism and nutrition disorders) | 113 | 43
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 16 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 12
Hypertension (Vascular disorders) | 60 | 20
Dysgeusia (Nervous system disorders) | 34 | 5
Headache (Nervous system disorders) | 19 | 11
Anaemia (Blood and lymphatic system disorders) | 77 | 52
Neutropenia (Blood and lymphatic system disorders) | 16 | 2
Urinary tract infection (Infections and infestations) | 35 | 21
COVID-19 (Infections and infestations) | 23 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 33
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 22 | 22
Proteinuria (Renal and urinary disorders) | 37 | 13
Haematuria (Renal and urinary disorders) | 18 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT04446117/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT04446117/SAP_001.pdf